CLINICAL TRIAL: NCT02004808
Title: Neutrophil Extracellular Traps and Sickle Cell Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: Tasmc-12-RE-0247-CTIL
Record Dates: First submitted 2013-10-15; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2012-07

CONDITIONS: Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 10CC of peripheral venous blood will be collected from each patient at several time points: at diagnosis ,during pain crisis , at Hydroxyurea treatment.
Oversight: Data Monitoring Committee: No

SUMMARY:
NETs formation in vaso-occlusive events in sickle cell disease and the role of hydroxyurea treatment.The study hypothesis is that NETs formation by neutrophils has a role in the induction of vaso occlusive disease in blood vessels. It is possible that high leukocyte count in children with sickle cell anemia is a bad prognostic sign due to NETs formation supporting occlusion of peripheral and central blood vessels.Hydroxyurea treatment might prevent vaso occlusive syndrome not only by increasing HbF but also by decreasing neutrophil count and inhibiting NETs formation.

ELIGIBILITY:
Inclusion Criteria:

* children who suffer from sickle cell disease and/or children with sickle cell disease treated with hydroxyurea

Exclusion Criteria:

* none

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Infants and children who suffer from sickle cell disease and/or Infants and children with sickle cell disease treated with hydroxyurea at the pediatric hemato-oncology department
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2014-02; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
measurements of neutrophil function | at first admition (day 1)

SECONDARY OUTCOMES:
measurements of neutrophil function | at sickle cell crisis while hospitalized

OTHER OUTCOMES:
measurements of neutrophil function | before and during treatment with hydroxyurea

CONTACTS AND LOCATIONS:
Overall Officials: Ronit Elhasid, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center